CLINICAL TRIAL: NCT01489891
Title: Usefulness of Applying Lidocaine as Topical Pharyngeal Anaesthesia in Esophagogastroduodenoscopies Performed Under Sedation With Propofol- a Randomized Controlled Trial
Brief Title: Usefulness of Lidocaine as Topical Pharyngeal Anaesthesia in Esophagogastroduodenoscopy Under Sedation With Propofol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Infanta Cristina (Other)
Responsible Party: Principal Investigator, Felipe de la Morena Lopez MD, Gastroenterologist. Head of endoscopy, Hospital Universitario Infanta Cristina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011-005704-15; ATF-EGD001
Record Dates: First submitted 2011-12-03; First posted 2011-12-12 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Esophagogastroduodenoscopy
Keywords: Esophagogastroduodenoscopy; Lidocaine; Propofol
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine group (Active Comparator): Blinded spraying 50 mg of pharyngeal topical lidocaine 180 seconds before sedated esophagogastroduodenoscopy (EGD)
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Excipients without lidocaine. The flavour taste is the same of active comparator ensuring the masking.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Applying of 5 puff controlled released (50 mg) transoral spray of lidocaine (10 mg=1 puff).
  Arms: Lidocaine group
Drug: Placebo — Applying of 5 puff controlled released (50 mg) transoral spray of placebo (excipients of trade mark of lidocaine ensuring the patient masking).
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of application of the anaesthesia topical pharyngeal with lidocaine in esophagogastroduodenoscopy under propofol´s sedation, in therms of dosage and side effect´s reduction overall.

ELIGIBILITY:
Inclusion Criteria:

* Patient´s over 18 years old that received standard indication for sedated esophagogastroduodenoscopy (American Society of Gastrointestinal Endoscopy Guidelines) in our centre between the period of study.

Exclusion Criteria:

* Patients under 18 years old
* Unable to obtain inform´s consent
* Emergency endoscopy
* Pregnant women
* Encephalopathy
* Well known allergic reaction to propofol, amide-anaesthesics, soy or eggs
* Methaemoglobinemia induced factor risks
* No previous or unknown fasting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe de la Morena, M.D., Principal Investigator
Locations (1):
- Hospital Universitario Infanta Cristina, Parla, Madrid, Spain

REFERENCES:
- [Result] Jimenez-Puente G, Hidalgo-Isla M. [Use of topical pharyngeal anaesthesia in esophagogastroduodenoscopy in unsedated patients]. Enferm Clin. 2011 Jan-Feb;21(1):30-4. doi: 10.1016/j.enfcli.2010.07.008. Epub 2011 Feb 18. Spanish. PMID 21334240
- [Result] Amornyotin S, Srikureja W, Chalayonnavin W, Kongphlay S, Chatchawankitkul S. Topical viscous lidocaine solution versus lidocaine spray for pharyngeal anesthesia in unsedated esophagogastroduodenoscopy. Endoscopy. 2009 Jul;41(7):581-6. doi: 10.1055/s-0029-1214865. Epub 2009 Jul 8. PMID 19588284
- [Result] Evans LT, Saberi S, Kim HM, Elta GH, Schoenfeld P. Pharyngeal anesthesia during sedated EGDs: is "the spray" beneficial? A meta-analysis and systematic review. Gastrointest Endosc. 2006 May;63(6):761-6. doi: 10.1016/j.gie.2005.11.059. PMID 16650534
- [Result] Lachter J, Jacobs R, Lavy A, Weisler A, Suissa A, Enat R, Eidelman S. Topical pharyngeal anesthesia for easing endoscopy: a double-blind, randomized, placebo-controlled study. Gastrointest Endosc. 1990 Jan-Feb;36(1):19-21. doi: 10.1016/s0016-5107(90)70915-7. PMID 2179038
- [Result] Mulcahy HE, Greaves RR, Ballinger A, Patchett SE, Riches A, Fairclough PD, Farthing MJ. A double-blind randomized trial of low-dose versus high-dose topical anaesthesia in unsedated upper gastrointestinal endoscopy. Aliment Pharmacol Ther. 1996 Dec;10(6):975-9. doi: 10.1046/j.1365-2036.1996.89261000.x. PMID 8971297
- [Result] Ristikankare M, Hartikainen J, Heikkinen M, Julkunen R. Is routine sedation or topical pharyngeal anesthesia beneficial during upper endoscopy? Gastrointest Endosc. 2004 Nov;60(5):686-94. doi: 10.1016/s0016-5107(04)02048-6. PMID 15557943
- [Result] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anaesthesiologist administration of propofol for GI endoscopy. Eur J Anaesthesiol. 2010 Dec;27(12):1016-30. doi: 10.1097/EJA.0b013e32834136bf. PMID 21068575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients over 18y with instructions for diagnostic or therapeutic EGD referred to the Endoscopy Unit of the Infanta Cristina Hospital for sedation were included successively. All patients was referred to the Infanta Cristina Hospital Endoscopy Unit in Parla, Madrid, Spain, for an EGD between January and May 2012.
Pre-assignment Details: The exclusion criteria were instructions for urgent endoscopy, encephalopathy, zero patient cooperation, lack of informed consent, not having fasted, a history to developing methemoglobinemia, pregnant women, lactating mothers or known allergies to propofol or lidocaine. All the patients provided their informed consent beforehand
Groups:
- Lidocaine Group: Blinded spraying 50 mg of pharyngeal topical lidocaine 180 seconds before sedated esophagogastroduodenoscopy (EGD)
  Lidocaine : Applying of 5 puff controlled released (50 mg) transoral spray of lidocaine (10 mg=1 puff).
- Placebo: Excipients without lidocaine. The flavour taste is the same of active comparator ensuring the masking.
  Placebo : Applying of 5 puff controlled released (50 mg) transoral spray of placebo (excipients of trade mark of lidocaine ensuring the patient masking).
Period: Overall Study
Arm/Group | Lidocaine Group | Placebo
Started | 60 | 60
Completed | 59 | 60
Not Completed | 1 | 0
Not completed — Endoscopy failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine Group: Blinded spraying 50 mg of pharyngeal topical lidocaine 180 seconds before sedated EGD
  Lidocaine : Applying of 5 puff controlled released (50 mg) transoral spray of lidocaine (10 mg=1 puff).
- Total: Total of all reporting groups
Arm/Group | Lidocaine Group | Placebo | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 46 | 93
  >=65 years | 12 | 14 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 49.7 (15.8) | 51.7 (14.9) | 50.7 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  Spain | 59 | 60 | 119

OUTCOME MEASURES:

1. Primary Outcome: Rate of Administration of Propofol 1% Required to Obtain Uniform Sedation During Endoscopy
Description: The propofol will be administered by an expert anaesthetist in repeated bolus (10-20 mg each 30-60 seconds) after an initial induction dosage (0.5-0.6 mg/kg ASA (American Society of Anaesthesiologists) I-II or 0.25-0.35 mg/kg ASA III-IV) to obtain an uniform level of sedation (OAAS 3 and bispectral index (BIS) 70-80) and adequate perceived patient tolerance (no gag-reflex, cough, sudden movements).
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: mcg/kg/min
Arm/Group | Lidocaine Group | Placebo
Number analyzed (Participants) | 59 | 60
mcg/kg/min | 310.7 (139.2) | 280.1 (87.7)
Statistical Analysis 1: Comparison: Lidocaine Group vs Placebo; Test type: Non-Inferiority or Equivalence — Beta 0.1; Alpha 0.05; p < 0.05, t-test, 2 sided; Median Difference (Final Values) = 30.6, Standard Deviation 42.1

2. Secondary Outcome: Percentage of Participants With Adverse Events in Both Groups
Description: Hypoxemia (SatO2<90% or >4% if the baseline was under 93%), bradycardia (<60 bpm or >10% from baseline), hypotension (systolic blood pressure under 90 mmHg and/or diastolic 60 mmHg), anaphylactic reaction, aspiration o methaemoglobinemia.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 hours postprocedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lidocaine Group | Placebo
Number analyzed (Participants) | 59 | 60
percentage of participants | 32.2 [21.6 to 45] | 26.7 [17 to 39]

3. Secondary Outcome: Likert Four Elements Scale to Evaluate the Satisfaction of Endoscopist
Description: Define as easiness to reach the expected objectives for endoscopy without patient interference: very satisfied, satisfied, neutral, unsatisfied.
Time Frame: 8 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lidocaine Group | Placebo
Number analyzed (Participants) | 59 | 60
percentage of participants
  Unsatisfactory | 6.8 [2.2 to 15.5] | 0 [0 to 4.8]
  Neutral | 10.1 [4.2 to 19.9] | 15 [7.6 to 25.7]
  Satisfactory | 25.4 [10 to 29.6] | 18.3 [15.5 to 37.6]
  Very satisfactory | 57.6 [54 to 77.7] | 66.6 [44.8 to 69.7]

4. Secondary Outcome: Likert Four Elements Scale to Evaluate the Satisfaction of Anaesthetist
Description: Define as easiness to reach and maintain the level of sedation and patient comfort during endoscopy: very satisfied, satisfied, neutral, unsatisfied.
Time Frame: 8 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lidocaine Group | Placebo
Number analyzed (Participants) | 59 | 60
percentage of participants
  Unsatisfactory | 5.8 [1.3 to 13.2] | 0 [0 to 4.8]
  Neutral | 16.9 [8.9 to 28.4] | 16.7 [8.8 to 27.7]
  Satisfactory | 15.2 [7.7 to 26.1] | 20.3 [11.3 to 31.6]
  Very satisfactory | 62.7 [49.9 to 74.3] | 63.3 [50.6 to 74.7]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Lidocaine Group | Placebo
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 19/59 | 16/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lidocaine Group (N=59) | Placebo (N=60)
Desaturation (Respiratory, thoracic and mediastinal disorders) | 11 | 9 — Desaturation is defined as in drop in SatO2<90% or >4% with respect to the basal figure if it were ≤93%.
Hypotension (Vascular disorders) | 12 | 11 — Hypotension is defined as a drop in systolic blood pressure < 90 mmHg or in diastolic blood pressure < 60 mmHg
Bradycardia (Cardiac disorders) | 2 | 4 — Bradycardia is defined as a <60 bmp drop in heart rate during the procedure or a >10% drop in relation to the basal figure

LIMITATIONS AND CAVEATS:
Unicenter study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No